CLINICAL TRIAL: NCT00949039
Title: Study Comparing Isolated Pelvic Perfusion With TNF-α 0.3 mg and Melphalan 1.5 mg/kg Versus Standard Treatment in Patients With Non Resectable, Recurrent Gynaecologic or Digestive Pelvic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIP2; CSET 1443
Record Dates: First submitted 2009-07-07; First posted 2009-07-30 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-03

CONDITIONS: Gynaecologic or Digestive Pelvic Cancer
MeSH Terms: interventions — Radiotherapy; Surgical Procedures, Operative

ARMS (2):
- Chemotherapy (Experimental): Isolated pelvis perfusion
  Interventions: Drug: Isolated pelvis perfusion
- Control (Active Comparator): Standard treatment
  Interventions: Radiation: radiotherapy; Procedure: Surgery

INTERVENTIONS:
Drug: Isolated pelvis perfusion — injection of TNF-α 0.3 mg followed 5 minutes later by melphalan 1,5mg/kg
  Arms: Chemotherapy
Radiation: radiotherapy — chemotherapy and/or radiotherapy and/or surgery
  Arms: Control
Procedure: Surgery
  Arms: Control

SUMMARY:
Randomised phase 3 trial comparing 2 arms: an experimental treatment (Isolated pelvis perfusion) and a standard treatment (systemic chemotherapy +/- radiotherapy +/- surgery).

Patients included have a non resectable, recurrent gynaecologic or digestive pelvic cancer.

The aim of the study is to show a 25% increase in 1 year overall survival rate with isolated pelvic perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proved locally advanced gynaecologic or digestive tumours (epidermoid carcinomas, adenocarcinomas, neuroendocrine tumours, sarcomas or melanomas), (cervix, vagina, rectal, anal).
* Locally recurrent tumours for which surgical treatment will be mutilating or marginal (R1 or R2) and/or for cervix cancer, primary tumours non accessible for standard treatment (radiotherapy- chemotherapy - brachytherapy and surgery).
* Surgically resectable tumour (R0 type) but for which patient does not agree with surgery.
* Patients aged over 18 and under 76 ans
* Performance OMS Index ≤ 2
* Normal biologic parameters
* Good general and cardiac state (ASA I or II and NYHA I or II)

Exclusion Criteria:

* Surgically resectable tumour (RO) or peritoneal tumour extension or distant metastasis.
* Cardiac or vascular pathology
* Pulmonary disease
* Uncontrolled Sepsis disease
* Pregnancy

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2009-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Survival rate | From randomization to death

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Gustave Roussy, Villejuif, France

REFERENCES:
- See also: Related Info — http://www.igr.fr/